CLINICAL TRIAL: NCT05024604
Title: Hysteroscopic Findings in Women Using Progesterone Only Pills (Minipills) Prospective Cohort Study .
Brief Title: Hysteroscopic Findings in Women Using Progesterone Only Pills (Minipills)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samuel Gendy (Other)
Responsible Party: Sponsor-Investigator, Samuel Gendy, Resident of Obstetrics & Gynecology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 117101333
Record Dates: First submitted 2021-08-04; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Women Health; Contraception
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: women receiving mini pills as a method of contraception with symptoms not diagnosed with us
  Interventions: Drug: Progesterone Only Product in Oral Dose Form; Other: office hysterscopy
- Control group: women attending to office hysteroscopy unit and not taking hormonal therapy
  Interventions: Other: office hysterscopy

INTERVENTIONS:
Drug: Progesterone Only Product in Oral Dose Form — mini pills as a contraceptive method
  Groups: study group
Other: office hysterscopy — office hysteroscoy

SUMMARY:
Hysteroscopic findings in women using progesterone only pills (minipills) :A Prospective cohort study.

DETAILED DESCRIPTION:
Hysteroscopic findings in women using progesterone only pills (minipills) :A Prospective cohort study. versus women not using any hormonal therapy ,Office hysteroscopy would be conducted outside of the formal operating theater setting in an appropriately sized, equipped, and staffed treatment room with adjoining, private changing facilities and toilet. As the patient is aware of everything that is going on, it is advisable to organize a relaxed setting, using a protected space with a comfortable seat, Uterine distension:

When performing diagnostic hysteroscopic procedures, it is best if a non-viscous, physiologic solution is used i.e. Saline or Lactated Ringers as opposed to CO2 gas. CO2 is commonly used for diagnostic hysteroscopy but is difficult to use in the presence of blood or mucous. Adequate distention pressures (50-70 mmHG) can be achieved in the office by the use of gravity or a pressure bags. Most office based procedures are of short duration and no more than 2 liters of solution should be utilized. In this situation, it is not necessary to monitor fluid inflow, outflow and deficits in the office setting. The standard access approach to the cervix involves placing a speculum within the vagina (preferably side opening), placing single tenaculum on the anterior lip of the cervix, injecting the cervix with local anaesthesia (if necessary), and placing the rigid continuous flow hysteroscope within the cervical canal. In most patients, including nulliparous and post menopausal patients, it is not necessary to dilate the cervix prior to insertion. Once the hysteroscope is within the cervical canal, the speculum should be removed, the fluid flow is begun and the hysteroscope is advanced through the cervical canal and into the uterine cavity under direct visualization.

The endometrium will be inspected by outpatient hysteroscopy The following observations made at hysteroscopy, and reviewed in detail from the video record of the examination Glandular and stromal changes The color, thickness, texture and regularity of the endometrial stroma would be assessed during hysteroscopy Superficial vascular density Endometrial vascular density would be assessed at hysteroscopy by direct inspection of the blood vessels, and graded according to the abundance of superficial vessels observed. Superficial vascular density would be reassessed after uterine collapse and Re distention.

Vascular morphology The shape and configuration of superficial and deep endometrial vessels would be assessed at hysteroscopy. The presence of regular and irregular (neo vascular and mosaic) vascular patterns in superficial and deep vessels would be recorded and graded. The presence of petechiae and ecchymosis would be recorded.

All the above values were regraded after collapse and re distention of the uterus, provided that a clear view of the endometrium could be obtained.

Vascular distribution The distribution of superficial and deep vasculature in the endometrium would be inspected and graded as even' or 'patchy'.

Endometrial biopsies biopsies would be taken at each hysteroscopy. A small amount of endometrial tissue was obtained under direct vision using the biopsy curette (novak curette). also a detailed comment by the examiner would be given regarding the uterine ostium of the fallopian tube & any changes in the cervical canal and the cervical secretions any abnormal findings or pathology would be mentioned also .

ELIGIBILITY:
Inclusion criteria:

* study group:

  * women using POP.
  * Age: reproductive age.
  * Symptoms: abnormal uterine bleeding without an organic cause.

    2-Authorization to participate in the study .
* Control group

  1- women attending to office hysteroscopy clinic
  * Age: reproductive Age
  * Contraception use : none.
  * Hormonal use: none.
  * Symptoms: abnormal uterine bleeding without an organic cause. All women in both groups would be subjected to Trans Vaginal U.S before doing hysteroscopy .

    b. Exclusion criteria:
* study group

  * Coagulopathies
  * Any contraindications to POPs as :
* past or current breast cancer, cirrhosis, and use of anticonvulsants
* suspected pregnancy
* current stroke or IHD
* severe hypertension

  •Any contraindications to hysteroscopy as :
* Pelvic infection
* Pregnancy
* Cervical cancer
* Heavy uterine bleeding.
* Control group --Women using any type of hormones including COCs .

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — reproducative age
Study Population: maternal health and family planning
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
primary outcome | an average of 1 year
  Hysteroscopic findings in women using POPs versus those not using hormones.( cervical mucosa , endometrium )

SECONDARY OUTCOMES:
subsidiary | an average of 1 year
  documentation of the local effects of POPs as a method of contraception

CONTACTS AND LOCATIONS:
Locations (1):
- Women health hospital , Assuit university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided